CLINICAL TRIAL: NCT01466140
Title: Effects of Writing Down the Request for Help With Regard to Patient Satisfaction in General Practices
Brief Title: Effects of Writing Down the Request for Help on Patient Satisfaction in General Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanne Kleefstra (Other)
Responsible Party: Sponsor-Investigator, Nanne Kleefstra, MD, PhD, assistant professor, Medical Research Foundation, The Netherlands
Organization: Medical Research Foundation, The Netherlands (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: EffectsPS1
Record Dates: First submitted 2011-10-21; First posted 2011-11-07 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-11

CONDITIONS: Patient Satisfaction; Doctor Satisfaction; Duration of Consultation
Keywords: Patient Satisfaction; Request for help; General practice
MeSH Terms: conditions — Patient Satisfaction | interventions — Insemination, Artificial, Heterologous

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Patients in the control group were asked to participate in a patient satisfaction study. They were asked to fill in a questionnaire with respect to patient satisfaction.
- Use of request card (Experimental): Patients in the intervention group were told that the practice was participating in a patient satisfaction study, and they were given an envelope with information about the 'doorknob phenomenon' and a request card. The envelope for the control group only consisted of information about a patient satisfaction study, without any information on the 'doorknob phenomenon', and without a request card. Both groups received the same letter with patient information about the study.
  Interventions: Other: Writing down request for help

INTERVENTIONS:
Other: Writing down request for help — Patients in the intervention group could write down their request for help on a request card (with a maximum of 2 questions).
  Arms: Use of request card

SUMMARY:
The primary objective of this study is to determine whether exploring the request for help more thoroughly improves patient satisfaction in general practice (primary care).

DETAILED DESCRIPTION:
Patient satisfaction has been an important topic of interest in primary health care during the last decade(s). Many factors during the consultation influence patient satisfaction. One of the aspects in a consultation is the request for help; especially in primary care the request for help has been recognised as an important aspect influencing patient satisfaction. The investigators hypothesized that exploring the request for help more thoroughly would improve patient satisfaction in general practice.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a new request for help.

Exclusion Criteria:

* Dementia
* Mental disability
* No or little knowledge of the Dutch language
* Illiteracy
* Limited vision

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction measured with the Consultation Satisfaction Questionnaire | 15-30 minutes (after the consultation patients filled in the questionnaire)
  The primary endpoint is the 'Professional Care' (PC) scale of the 'Consultation Satisfaction Questionnaire' (CSQ). In a previous study the score on the PC were 88.2 en 80.9 in the intervention and control groups, respectively. The standard deviations were 11.8 en 16.1. For our sample size calculation we used an expected standard deviation of 15. The sample size required to detect a difference of 7 on the PC scale between the intervention and control group, with a power of 90%, and alpha of 5% (two-tailed), and a standard deviation of 15, was 196 patients. We rounded this number off to 200.

SECONDARY OUTCOMES:
Patient satisfaction measured with the Visual Analog Scale | 15-30 minutes (patients filled in the Visual Analog Scale after the consultation)
  On a scale of 0-10 patients could fill in the Visual Analog Scale with regard to the patient satisfaction during the consultation
Doctor satisfaction measured with the Visual Analog Scale | 15-30 minutes (general pracitioners filled in the Visual Analog Scale after the consultation)
  On a scale from 0-10 general practitioners could fill in the Visual Analog Scale with regard to their own satisfaction about the consultation
Duration of the consultation | 15-30 minutes (after the consultation the doctor measured the time with a stopwatch)
  Duration of the consultation was compared between both groups

CONTACTS AND LOCATIONS:
Overall Officials: Henk Bilo, Study Chair — Medical Research Centre
Locations (1):
- Isala Clinics, Zwolle, Overijssel, Netherlands